CLINICAL TRIAL: NCT04736589
Title: Efficacy and Safety of Inetetamab Combined With Rapamycin and Chemotherapy for HER2-positive Metastatic Breast Cancer Patients With Abnormal Activation of PI3K/Akt/mTOR Pathway After Progression on Trastuzumab.
Brief Title: Inetetamab Plus Rapamycin and Chemotherapy for HER2+ Metastatic Breast Cancer With Abnormal Activation of PAM Pathway
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Fei Ma, Associate director of the department of Medical Oncology in Cancer Hospital，Chinese Academy of Medical Sciences and Peking Union Medical College, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR-1.1
Record Dates: First submitted 2021-01-31; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Inetetamab; Rapamycin; PI3K/Akt/mTOR pathway
MeSH Terms: conditions — Breast Neoplasms | interventions — Sirolimus; pyrotinib; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inetetamab plus Rapamycin plus Chemotherapy (Experimental): Drug: Inetetamab Initial dose of 8mg/kg, completed in 90 minutes IV infusion, and then 6 mg/kg over 30-90 minutes IV infusion every 3 weeks, until disease progression (PD) or other termination criteria are met;
  Drug: Rapamycin Oral 2mg, once a day;
  Drug: Chemotherapy drugs are not limited in this trial, please refer to their instructions for specific usage.
  Interventions: Drug: Inetetamab; Drug: Rapamycin; Drug: Chemotherapy
- Pyrotinib plus chemotherapy (Active Comparator): Drug:Pyrotinib Oral 400mg, once a day;
  Drug: Chemotherapy drugs are not limited in this trial, please refer to their instructions for specific usage.
  Interventions: Drug: Pyrotinib; Drug: Chemotherapy

INTERVENTIONS:
Drug: Inetetamab — Initial dose of 8mg/kg, completed in 90 minutes IV infusion, and then 6 mg/kg over 30-90 minutes IV infusion every 3 weeks.
  Arms: Inetetamab plus Rapamycin plus Chemotherapy
Drug: Rapamycin — Oral 2mg, once a day.
  Arms: Inetetamab plus Rapamycin plus Chemotherapy
Drug: Pyrotinib — Oral 400mg, once a day.
  Arms: Pyrotinib plus chemotherapy
Drug: Chemotherapy — Chemotherapy drugs are not limited in this trial, please refer to their instructions for specific usage.

SUMMARY:
This is a multi-center,randomized,phase 3 clinical trial. In the study, HER2-positive metastatic breast cancer patients with abnormal activation of PI3K/Akt/mTOR pathway after progression on trastuzumab are enrolled and randomized to receive the treatment of Inetetamab plus Rapamycin plus chemotherapy or Pyrotinib plus chemotherapy.The study aimed to access the efficacy and safety of Inetetamab combined with Rapamycin and chemotherapy in HER2-positive metastatic breast cancer patients with abnormal activation of PI3K/Akt/mTOR pathway.

DETAILED DESCRIPTION:
This is a multi-center,randomized,phase 3 clinical trial. In the study, HER2-positive metastatic breast cancer patients with abnormal activation of PI3K/Akt/mTOR pathway after progression on trastuzumab are enrolled and randomized to receive the treatment of Inetetamab plus Rapamycin plus chemotherapy or Pyrotinib plus chemotherapy.The study aimed to access the efficacy and safety of Inetetamab combined with Rapamycin and chemotherapy in HER2-positive metastatic breast cancer patients with abnormal activation of PI3K/Akt/mTOR pathway after progression on trastuzumab. The primary end point is Progressive-free Survival (PFS). The secondary end points are Overall Response Rate (ORR),Overall Survival (OS),Clinical Benefit Rate (CBR) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Female, Aged > 18;
2. HER2-positive breast cancer are defined as immunohistochemical (IHC) testing as +++, or IHC++ with FISH testing of positive;
3. Histologically or cytologically confirmed invasive breast carcinoma with locally recurrent or radiological evidence of metastatic disease.
4. Patients with HER2-positive metastatic breast cancer who have progressed disease after trastuzumab treatment include the following four types of patients (Note: The following patients are in a parallel relationship):

   1. Patients with HER2-positive breast cancer who have progressed during adjuvant trastuzumab treatment after surgery; or
   2. Patients with HER2-positive breast cancer who have relapsed or metastasized after receiving adjuvant trastuzumab therapy; or
   3. HER2-positive recurrent or metastatic BC patients who have progressed after receiving at least 4 weeks of trastuzumab as first-line treatment ; or
   4. HER2-positive metastatic BC patients who have never been treated have progressed after receiving at least 4 weeks of trastuzumab as first-line treatment.
5. Genetic testing shows that the PI3K/Akt/mTOR pathway related genes are mutated;
6. ECOG PS score ≤2, estimated survival time ≥6 months, and can be followed-up;
7. Patients with measurable disease as per RECIST 1.1 criteria;
8. Cardiopulmonary function is basically normal, LVEF≥50% within 4 weeks before starting treatment;
9. An adequate liver function with the following definition:

   1. Total bilirubin ≤ 1.5 times the upper limit of normal value. Patients with known Gibert's disease can be included in the group if combined bilirubin ≤ 1.5 times the upper limit of normal value;
   2. AST and ALT ≤2.5 times the upper limit of the normal value; if there is liver metastasis, ≤5 times the upper limit of the normal value (the normal value is the normal value specified by this clinical trial center);
10. Have sufficient baseline hematology parameters, defined as follows:

    1. ANC≥1.5 x 10^3 /μL;
    2. Platelet count ≥100 x 10^3/μL, if it is 75-100 x 10^3/μL, it may be included in the group, as long as the doctors believe it can be included;
    3. Hemoglobin ≥9 g/dL.
11. Coagulation Indicators: International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 times the upper limit of normal, unless drugs known to change INR and aPTT are used;
12. No history of serious heart, kidney and other important organs and endocrine disease;
13. Female patients of childbearing age have a negative pregnancy test and voluntarily take effective and reliable contraceptive measures;
14. The patients voluntarily signed an informed consent form.

Exclusion Criteria:

Anyone who has one of the following conditions cannot be selected for this trial:

1. Participated in other clinical trials within 4 weeks;
2. Have used mTOR inhibitors in the past;
3. Previous use of Pyrotinib in first-line treatment stage; previous use of lapatinib is allowed;
4. Accompanied by immunosuppressant or chronic corticosteroid medication, or more than 25% bone marrow radiotherapy within 4 weeks;
5. Symptomatic CNS metastases or evidence of leptomeningeal disease;
6. Gastrointestinal dysfunction or gastrointestinal diseases (including active ulcers);
7. Hepatitis B or hepatitis C carriers, or other known chronic liver diseases; HIV positive;
8. Known hypersensitivity to any study medication
9. Women during pregnancy or lactation;
10. Left ventricular ejection fraction <50%; clinical manifestations of patients with obvious arrhythmia, myocardial ischemia, severe atrioventricular block, cardiac insufficiency, and severe valvular disease;
11. Any malignancy within 5 years prior to randomization, with the exception of adequately treated in-situ carcinoma of the cervix uteri, basal or squamous cell carcinoma;
12. The researchers decide that any other medical, social or psychological conditions which are inappropriate to participate in this trial.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-02-02 (Estimated); Primary Completion 2024-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Progressive-free Survival (PFS) | Estimated 24 months
  Progressive-free Survival (PFS) is defined as the time from the date of randomization to the date of first radiologically documented tumor progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Estimated 24 months
  Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Overall Survival （OS） | Estimated 48 months
  Overall Survival （OS）is defined as the time from date of randomization to the date of death from any cause.
Clinical Benefit Rate (CBR) | Estimated 24 months
  Clinical Benefit Rate (CBR) is defined as the percentage of participants whose best overall response, according to RECIST1.1, is either complete response (CR), a partial response (PR) or stable disease (SD) lasting for at least 24 weeks.
Safety(AEs and SAEs) | From consent through 28 days following treatment completion
  Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China